CLINICAL TRIAL: NCT02988193
Title: Piloting Healthcare Coordination in Hypertension
Acronym: PRECISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Optima Integrated Health (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-16045
Record Dates: First submitted 2016-12-02; First posted 2016-12-09 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-03

CONDITIONS: Hypertension
Keywords: clinical reasoning artificial intelligence; poorly controlled hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The medication treatment intervention between arms differs in that the optima4BP arm uses an analytic intelligence algorithm to optimize drug treatment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- optima4BP Medication Management (Experimental): optima4BP will provide a monthly medication optimization to the treating physician for review and subsequent implementation. The Treatment Recommendation will consist of:
  1. curated blood pressure (BP) and heart rate (HR) values reported by the patient through the use of home monitoring BP arm cuff;
  2. medication treatment recommendation;
  3. active link to access additional treatment analysis tools.
  Interventions: Device: optima4BP Medication Management
- Usual Care Medication Management (No Intervention): Usual care management will follow medication treatment management according to the physician preference. The treating physician will not be provided with a medication optimization recommendation, nor with monthly curated BP and HR values.

INTERVENTIONS:
Device: optima4BP Medication Management — A clinical reasoning expert system is used to determine the need for a medication treatment optimization. If a treatment optimization is needed, the expert system generates a recommendation that is sent to the treating physician.
  Arms: optima4BP Medication Management

SUMMARY:
The PRECISION study investigates the possibility of integrating a clinical decision support analytic intelligence into the clinical care flow at University of California San Francisco Medical Center (UCSF MC). optima-for-blood pressure [optima4BP], our innovation, transforms the episodic and reactive nature of uncontrolled HTN pharmacological treatment management into a process that is continuous, proactive, and personalized.

In addition, the clinical adoption of this "technology of the future" will be investigated to establish its feasibility in being embedded into the clinical care flow.

Today's hypertension (HTN) management paradigm often fails to align current patient health status with the most effective medication treatment. Without surveillance and rapid-cycles analysis of current patient health status and treatment efficacy, HTN management remains a struggle. optima4BP addresses pharmacological intervention management by identifying the need for a drug treatment change and recommending the most appropriate drug optimization.

The PRECISION study represent a pilot trial intended to address 2 critical design components of optima4BP:

1. Can optima4BP interoperate with multiple IT platforms to collect and distribute data?
2. What is the treating physician confidence in using optima4BP?

DETAILED DESCRIPTION:
Goal: Conduct a prospective randomized pilot clinical trial embedded within the care delivery system at UCSF Medical Center (UCSF). It is intended to evaluate the efficacy of optima4BP in improving care coordination for patients with uncontrolled hypertension (HTN). Although optima4BP has been evaluated during patient-physician office visits, it has not been evaluated for its efficacy to support treatment changes remotely, over time. PRECISION investigates this aspect and its impact on stakeholders (physicians and patients). The outcomes will set the stage for a scaled-up study of 300 patients at UCSF.

Study Design: The patients will be randomized to 2 arms (a) optima4BP surveillance and treatment recommendation support (O4BP); (b) usual care (UC) - usual care seen appropriate by the treating physician). NOTE: The original design prior to study initiation considered a 3 arms randomization which would also include: enhanced care (EC) representing a "step up" from UC by providing the physician with raw remotely collected BP values sent on a monthly cycle. However, this arm was abandoned at enrollment because patients in the UC arm were proactively reaching out to their physicians with remotely collected BP values from the Qardio® device therefore rendering the initially projected Extended Care arm unuseful.

Every 30 days, the collection of patient information will be followed by an arm-specific action. For identified patients in need of a medication change, O4BP physicians will receive a treatment change recommendation for review. UC physicians will not receive any information. All patients will undergo at least 2 in-office visits, a baseline visit and an exit visit. All patients will be asked to provide every 30 days the following information: (a) adherence to current HTN treatment; and (b) experienced side-effects and severity. The communication will be performed via e-mail between Health-e-Heart (HeH) automated system (https://www.health-eheartstudy.org/) and the patient. HeH will automatically obtain BP values from the remote monitors provided to each patient.

ELIGIBILITY:
Inclusion Criteria:

* UCSF General Medicine patient
* 2 or more values on consecutive office visits within 12 months: systolic blood pressure (SBP) > 140 mmHg or diastolic blood pressure (DBP) > 90
* Therapy with at least 2 anti-hypertensive pharmacological classes at the time of the last office visit

Exclusion Criteria:

* Does not own a smartphone
* Does not speak or read English
* Planning to leave UCSF in the next year
* Has a treating physician who refuses to enroll patients
* Treating physician states that:

Patient cannot manage Qardio® arm blood pressure (BP) device (due to cognitive, psychological, physical or other problems), or Patient is already at goal, or Should not participate in the study for any other reason

* Non-compliance with medical follow-up (frequent "no shows")
* Planned coronary revascularization in the next 6 months
* Myocardial infarction, stroke, coronary revascularization, cardiac or aortic surgery in the last 3 months

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela Voskerician, PhD, Principal Investigator — Optima Integrated Health; Liviu Klein, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Carlos, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- optima4BP Medication Optimization: optima4BP will provide a monthly medication optimization to the treating physician for review and subsequent implementation. The Treatment Recommendation will consist of:
  1. curated blood pressure (BP) and heart rate (HR) values reported by the patient through the use of home monitoring BP arm cuff;
  2. medication treatment recommendation;
  3. active link to access additional analysis tools.
  optima4BP medication optimization: A clinical reasoning expert system is used to determine the need for a medication treatment optimization. If a treatment optimization is needed, the expert system generates a recommendation that is sent to the treating physician.
- Usual Care Management: Usual care management will follow medication treatment management according to the physician preference. The treating physician will not be provided with a medication optimization recommendation, nor with monthly curated BP and HR values.
Period: Overall Study
Arm/Group | optima4BP Medication Optimization | Usual Care Management
Started | 12 | 16
Completed | 12 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- optima4BP Medication Management: optima4BP will provide a monthly medication optimization to the treating physician for review and subsequent implementation. The Treatment Recommendation will consist of:
  1. curated blood pressure (BP) and heart rate (HR) values reported by the patient through the use of home monitoring BP arm cuff;
  2. medication treatment recommendation;
  3. active link to access additional analysis tools.
  optima4BP Medication Management: A clinical reasoning expert system is used to determine the need for a medication treatment optimization. If a treatment optimization is needed, the expert system generates a recommendation that is sent to the treating physician.
- Usual Care Medication Management: Usual Care Medication Management will follow medication treatment management according to the physician preference. The treating physician will not be provided with a medication optimization recommendation, nor with monthly curated BP and HR values.
- Total: Total of all reporting groups
Arm/Group | optima4BP Medication Management | Usual Care Medication Management | Total
Number analyzed (Participants) | 12 | 16 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 12 | 16 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (3) | 69 (5) | 70 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 5 | 10 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 16 | 28

OUTCOME MEASURES:

1. Primary Outcome: Clinical Adoption of a Decision Support Artificial Intelligence
Description: Total number of participants that undergone a treatment change.
  This measure allows to evaluate the adoption of the optima4BP treatment recommendation based on the total number of patients that benefited from a treatment recommendation that was implemented by the treating physician.
Time Frame: 6 months
Population: Clinical adoption based on physician acceptance of the treatment recommendation
Measure: Count of Participants; unit: Participants
Groups:
- optima4BP Treatment Management: optima4BP will provide a monthly medication optimization to the treating physician for review and subsequent implementation. The Treatment Recommendation will consist of:
  1. curated blood pressure (BP) and heart rate (HR) values reported by the patient through the use of home monitoring BP arm cuff;
  2. medication treatment recommendation;
  3. active link to access additional analysis tools.
  optima4BP medication optimization: A clinical reasoning expert system is used to determine the need for a medication treatment optimization. If a treatment optimization is needed, the expert system generates a recommendation that is sent to the treating physician.
- Usual Care Treatment Management: Usual care management will follow medication treatment management according to the physician preference. The treating physician will not be provided with a medication optimization recommendation, nor with monthly curated BP and HR values.
Arm/Group | optima4BP Treatment Management | Usual Care Treatment Management
Number analyzed (Participants) | 12 | 16
Participants | 10 | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire course of the 6 months study.
Description: The definition of adverse event does not differ from clinicaltrials.gov Definition.
Arm/Group | optima4BP Treatment Management | Usual Care Treatment Management
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/16
Other Adverse Events (participants affected / at risk) | 0/12 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No